CLINICAL TRIAL: NCT05111275
Title: Impact of Cognitive Exercises on Cognitive Disorders in Survivors of a Prolonged ICU Stay.
Brief Title: Cognitive Exercises in Survivors of a Prolonged ICU Stay.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Anne-Françoise Rousseau, Head of Clinic, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MEMO
Record Dates: First submitted 2021-10-30; First posted 2021-11-08 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Critical Illness; Cognition Disorder
MeSH Terms: conditions — Critical Illness; Cognition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group MEMO (Experimental): Patients will perform cognitive exercises on the MEMO site at least 4 times per week for a month. During this month, patients will be contacted by phone on a weekly basis in order to maintain their motivation and ensure their treatment compliance. The time spent on the site during the month of evaluation will be quantified by the study investigator, via the professional profile created on the MEMO site, allowing to see the patient's activity on this same site.
  Interventions: Other: Cognitive exercises
- Control Group (No Intervention): Patients will not change their habits or perform cognitive exercises during the same assessment period.

INTERVENTIONS:
Other: Cognitive exercises — Exercises that stimulate and train memory, attention, executive functions, language and gnosis.
  Arms: Group MEMO

SUMMARY:
This study concerns patients who survived intensive care, after a minimum stay of 7 days and presenting cognitive disorders (with a score ≤ 26 on the MoCA test) during the post-intensive care follow-up consultation one month after ICU discharge.

The objective of this prospective open-label randomized study is to assess the impact of cognitive stimulation on recovery from cognitive impairment after a critical illness.

DETAILED DESCRIPTION:
Patients who survive a critical illness and a stay in intensive care may present a post-intensive care syndrome. This syndrome comprises in particular cognitive disorders, with memory disorders and executive disorders. The systemic inflammatory reaction seems to play an important role in the genesis of these disorders. Frequently reported risk factors are numerous and include hypoxemia, hypotension, glycemic dysregulation, drug toxicities, and, delirium.

In post-intensive care, these cognitive disorders are most often detected using screening tests that quickly and superficially assess the major components of cognition. During the standardized screening that we offer to patients who join the follow-up clinic of our university hospital, we use the MoCA (Montreal Cognitive Assessment) as a screening test. In a series of patients who survived a severe form of COVID-19, we observed that more than 80% of patients did not achieve the maximum score on this test (MoCA <30/30) 3 months after ICU discharge, thus signifying the presence of cognitive impairment. Half of these patients had mild disorders (MoCA> 26/30), the other half had more pronounced disorders, based on commonly accepted cut-off values (MoCA ≤ 26/30). Similar data are reported in other populations: cognitive disorders are frequently encountered after ARDS of other etiologies [5, 6], and may persist for several years after the acute episode [7].

In Belgium, access to an exhaustive cognitive assessment and cognitive rehabilitation is subject to different access criteria, which are not necessarily met by patients who have survived intensive care. Such rehabilitation is then quite expensive for the patient. Patients with cognitive impairment after intensive care may nevertheless benefit from aids in cognitive recovery. In a few rare studies, it seems that non-specific cognitive training can improve the cognitive outcome of patients who have survived intensive care [8].

According to several neuropsychologists interviewed as part of a preliminary investigation, there are cognitive stimulation tools that could activate spontaneous cognitive recovery in post-intensive care. Among them, the MEMO website (http://www.memory-motivation.org/home-2/) offers free access to batteries of cognitive exercises. This website was created by a team of psychologists, doctors, engineers and researchers in connection with the University of Nice Sophia Antipolis. It was designed to meet the needs of patients with cognitive disorders, healthcare professionals involved in prevention, rehabilitation and cognitive stimulation. This computer hardware playfully stimulates memory, attention, executive functions, language and gnosias. Several levels of difficulty are foreseen. In addition, the prescriber, by creating a professional profile on the website, can monitor the compliance and performance of patients to whom he has advised this platform.

This tool is intended as a means of stimulating cognitive recovery, but does not replace neuropsychological management in the event of persistent cognitive disorders.

The aim of our prospective randomized study is to assess the impact of cognitive stimulation on the course of cognitive impairment within two months of discharge from intensive care. Cognitive exercise cannot be offered too soon after the critical episode because patients are extremely tired. On the contrary, these exercises cannot be postponed too long in order to optimize the recovery as quickly as possible to the best possible functional state.

ELIGIBILITY:
Inclusion Criteria:

* Survivor of an ICU stay of at least 7 days
* Score ≤ 26 at the MoCA test at inclusion
* French speaker

Exclusion Criteria:

* Blindness
* Known mental disability
* Known dementia
* Cognitive rehabilitation in progress
* No internet connection
* Patient not knowing how to use the internet
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive disorders | At one month after inclusion
  Cognitive disorders assessed by the MoCA (Montreal Cognitive Assessment) test
Cognitive disorders | At one month after inclusion
  Cognitive disorders assessed by the RBANS (Repeatable Battery for the Assessment of Neuropsychological Status) test

OTHER OUTCOMES:
Cognitive activities | At one month after inclusion
  Quantification of the time dedicated to cognitive tasks during ICU stay (i.e.: reading, playing, cooking)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No